CLINICAL TRIAL: NCT01095302
Title: An Open-label, Dose-escalation, Safety and Pharmacokinetics Phase I Study of Ombrabulin in Combination With Docetaxel and Cisplatin Every 3 Weeks in Patients With Advanced Solid Tumors
Brief Title: Dose Escalation, Safety and Pharmacokinetic Study of AVE8062 Combined With Docetaxel and Cisplatin in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11089; U1111-1116-5905 (Other: UTN)
Record Dates: First submitted 2010-03-23; First posted 2010-03-30 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Neoplasms, Malignant
MeSH Terms: conditions — Neoplasms | interventions — AC 7700; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ombrabulin/ docetaxel/cisplatin (Experimental): AVE8062 combined with docetaxel and cisplatin will be administered once in every 3 weeks, with 30-minute intravenous infusion
  Interventions: Drug: OMBRABULIN (AVE8062); Drug: cisplatin; Drug: docetaxel

INTERVENTIONS:
Drug: OMBRABULIN (AVE8062) — Pharmaceutical form:injection solution
  Route of administration: intravenous infusion
Drug: cisplatin — Pharmaceutical form:injection solution
  Route of administration: intravenous infusion
Drug: docetaxel — Pharmaceutical form:injection solution
  Route of administration: intravenous infusion

SUMMARY:
Primary Objective:

* To determine the maximum tolerated dose based on the incidence of dose limiting toxicity and the maximum administered dose of ombrabulin in combination with docetaxel and cisplatin administered every 3 weeks in patients with advanced solid tumors

Secondary Objectives:

* To assess the overall safety profile of the combination therapy
* To characterize the pharmacokinetic profile of ombrabulin, its active metabolite RPR 258063, docetaxel and cisplatin in combination.
* To evaluate anti-tumor activity of the combination therapy

DETAILED DESCRIPTION:
The duration of the study for each patient will include an up to 4-week screening phase, 21-day study treatment cycles, an end of treatment visit and a follow-up period 30 days after the last infusion of ombrabulin. The patient will continue treatment until disease progression, unacceptable toxicity, patient's refusal of further treatment.

ELIGIBILITY:
Inclusion criteria:

* Patients with advanced solid tumor for which docetaxel and cisplatin is approved such as lung cancer, epithelial ovarian cancer.

Exclusion criteria:

* Eastern Cooperative Oncology Group performance status > or = 2.
* Concurrent treatment with any other anticancer therapy.
* Male or female patients who do not agree with contraception.
* Washout period of less than 28 days from prior anticancer therapies (chemotherapy, targeted agents, immunotherapy and radiotherapy) or any investigational treatment, except for nitrosoureas, mitomycin which may not be used up to 42 days prior to the first cycle. No washout period is required for hormonal therapy that has to be discontinued before the first cycle.
* Not recovered from all previous therapies (radiation, surgery, and medications). Adverse events related to previous therapies must be National Cancer Institute Common Terminology Criteria (NCI-CTCAE V3.0) grade < or = 1 (or alopecia < or = grade 2) at screening or returned to the subject's baseline prior to their most recent previous therapy.
* Symptomatic brain metastases and carcinomatous leptomeningitis.
* Other serious illness or medical conditions not controlled by adequate treatment
* Patients with more than 1 line of previous chemotherapy for advanced or metastatic disease (adjuvant/neoadjuvant and targeted agents [eg gefitinib] excluded).
* Current peripheral neuropathy > or = grade 2 and ototoxicity, of any origin including significant residual symptoms due to the use of neurotoxic drugs (eg vincaalkaloids, platinum and taxanes).
* Inadequate organ function
* Documented medical history of myocardial infarction, documented angina pectoris, arrhythmia especially severe conduction disorder such as second or third degree atrio-ventricular block, stroke, or history of arterial or venous thrombo-embolism within the past 180 days requiring anticoagulants.
* Patient with a left ventricular ejection fraction <50% by echocardiography.
* Patients with a baseline QTc interval >0.45, or family history of Long QT Syndrome.
* Patient with uncontrolled hypertension and patient with organ damage related to hypertension such as left ventricular hypertrophy or grade 2 ocular fundoscopic changes or kidney impairment.
* Patients with growing vessel disease (eg age-related macular degeneration, diabetic retinopathy, rheumatoid arthritis), or ongoing wound healing process. Patients should be enrolled in the study at least 28 days after surgery.
* 12-lead Electrocardiogram: ST- and T-wave changes suggesting ischemia
* Hypertension defined as systolic blood pressure (BP)>140 mmHg or diastolic BP>90 mmHg on two repeated measurements at 30 minutes intervals.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 3 weeks (cycle 1)

SECONDARY OUTCOMES:
Global safety profile based on treatment emergent adverse events, serious adverse events, and laboratory abnormalities | on-treatment period + 30 days
Pharmacokinetic profiles of all study drugs and AVE8062 active metabolite based on PK parameters (Cmax, AUC, t1/2, CL, Vss). | Cycle 1: Day 1 and 3; up to Cycle 4: Day 1
Objective tumor response as defined by the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | on-treatment period + 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Japan (3):
  - Investigational Site Number 392003, Akashi-Shi
  - Investigational Site Number 392001, Kōtoku
  - Investigational Site Number 392002, Nagoya

REFERENCES:
- [Derived] Nishio M, Satouchi M, Horiike A, Horio Y, Sunaga Y, Ecstein-Fraisse E, Hida T. Phase 1 study of ombrabulin in combination with docetaxel and cisplatin in Japanese patients with advanced solid tumors. Jpn J Clin Oncol. 2018 Apr 1;48(4):322-328. doi: 10.1093/jjco/hyy026. PMID 29514256